CLINICAL TRIAL: NCT00763633
Title: Vitamin B6 Concentration and Treatment in Nausea and Vomiting of Pregnancy
Brief Title: B6 Treatment for Nausea and Vomiting in Pregnancy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Showa University (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Dept. Obstetrics Gynecology Fac. Medicine Univ. Indonesia, Univ. Indonesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B601
Record Dates: First submitted 2008-09-29; First posted 2008-10-01 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-09

CONDITIONS: Nausea and Vomiting Complain in Early Pregnancy
Keywords: nausea; vomiting; pregnancy; B6
MeSH Terms: conditions — Nausea; Vomiting | interventions — Vitamin B 6

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- highB6 (Active Comparator): high vitamin B6
  Interventions: Drug: vitamin B6
- lowB6 (Active Comparator): low vitamin B6
  Interventions: Drug: vitamin B6

INTERVENTIONS:
Drug: vitamin B6 — high dose of vitamin B6
  Arms: highB6
Drug: vitamin B6 — low vitamin B6
  Arms: lowB6

SUMMARY:
The purpose of this study is to determine vitamin B6 concentration and whether vitamin B6 is effective in nausea and vomiting of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Nausea and vomiting of pregnancy

Exclusion Criteria:

* Other medical condition causing nausea and vomiting of pregnancy

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Nausea and vomiting score | 2 weeks

SECONDARY OUTCOMES:
Vitamin B6 concentration in nausea and vomiting of pregnancy | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Noroyono Wibowo, MD, PhD, Principal Investigator — Dept. Obstetric Gynecology Univ. Indonesia
Locations (1):
- Dept. Obstetric Gynecology Univ. Indonesia, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- See also: Univ. Indonesia web-link — http://www.ui.ac.id/en